CLINICAL TRIAL: NCT01072799
Title: A Phase 2 Study to Assess the Safety and Immunogenicity of an A (H1N1) 2009 Influenza Virus-like Particle (VLP) Vaccine
Brief Title: Safety and Immunogenicity of an A (H1N1) 2009 Influenza Virus-like Particle (VLP) Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NVX 754 H1N1-MEX
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Seasonal Influenza
Keywords: A (H1N1)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose H1N1 (Experimental)
  Interventions: Biological: A/H1N1 2009 Influenza VLP Vaccine
- Mid dose H1N1 (Experimental)
  Interventions: Biological: A/H1N1 2009 Influenza VLP Vaccine
- High dose H1N1 (Experimental)
  Interventions: Biological: A/H1N1 2009 Influenza VLP Vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Two doses (Day 1 and Day 22); 0.5mL
  Arms: Placebo
Biological: A/H1N1 2009 Influenza VLP Vaccine — Two doses (Day 1 & Day 22); 0.5mL
  Arms: High dose H1N1; Low dose H1N1; Mid dose H1N1

SUMMARY:
This is a Phase 2 randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability and immunogenicity of three dose levels (5µg, 15µg and 45µg HA) of the novel A (H1N1) influenza VLP vaccine as compared with a placebo in healthy adults (18 to 64 years of age).

DETAILED DESCRIPTION:
The study will be conducted in two parts (A & B) at a single center in Mexico. The purpose of Part A is to evaluate the safety of the H1N1 VLP vaccine and to evaluate immunogenicity and select a dose for Part B. In Part A, 1,000 subjects will be enrolled and randomized to a 1:1:1:1 schedule (5µg, 15µg and 45µg doses of H1N1 VLP vaccine or placebo. Subjects will receive two intramuscular (IM) injections (0.5mL/dose) of the H1N1 VLP vaccine or placebo 21 days apart. Blood for HAI assays will be collected at 3 time points (baseline, Day 14 and Day 36). Subjects will be followed for all adverse events (AEs) from the first day of the study through 21 days after the second dose (Day 36). Subjects will be followed for serious AEs and significant new medical conditions (SNMCs) to the end of the study 6 months post-dose 2 (Day 194).

Once the first 500 subjects are enrolled into Part A, enrollment will be halted until 3 days of safety follow-up data are reviewed by the study Data and Safety Monitoring Board (DSMB). A second data review will occur following Day 14 visit for Part A to select the dose to be administered in Part B.

Part B of the study will be conducted to evaluate safety and accumulate enough safety data to potentially move forward with broader use of the vaccine assuming favorable results. In Part B, a total of 3,250 - 3,750 subjects will be randomized to receive the selected dose of H1N1 VLP vaccine or placebo. A total of 3,000 H1N1 VLP vaccine recipients at the selected dose or higher, and 1,250 placebo recipients will be enrolled in Parts A and B. Following completion of Day 36 in Part A, data may be reviewed to assess 1 injection vs. 2 injections in Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-64 years of age at the time of the vaccination.
2. Informed consent must be obtained from the subject prior to beginning any study specific procedures indicating that they understand the purpose of this study and are willing to adhere to the procedures described in this protocol.
3. Available by telephone.
4. Free of obvious health problems or chronic illnesses (e.g., recent exacerbation or acute episode of chronic illness in the last 3 months) as established by medical history, review of systems, and clinical examination before entering the study. This includes any mental condition that would interfere with subject self-assessment. Subjects with a pre-existing chronic disease will be allowed to participate if the disease is stable. Stable disease is defined as no new onset of exacerbation of pre-existing chronic disease 3 months prior to study vaccine injection.
5. Female of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (e.g., intrauterine contraceptive device; oral contraceptives or other equivalent hormonal contraception) for 2 months prior to vaccination. Subject must also have a negative pregnancy test at study entry then at Day 22 and must agree to continue to use adequate contraceptive precautions for three months after vaccination.

Exclusion Criteria:

1. Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
2. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study (prior to the Day 201 follow-up call - 180 days after the second vaccination).
3. Have received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following the second vaccination.
4. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. The use of topical, inhaled and nasal steroids will be permitted.
5. Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
6. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
7. Acute disease on the day of vaccination (baseline/dose 1 or dose 2). Acute disease is defined as the presence of a moderate or severe illness with or without fever > 38 C.
8. Acute clinically-significant pulmonary (including asthma), cardiovascular, hepatic or renal functional abnormality as determined by physical examination or laboratory screening tests.
9. Major congenital defects that may increase the risk for complications from influenza.
10. History of any neurological disorders or seizures (with the exception of febrile seizures during childhood) related to an underlying immune disease or disorder, such as but not limited to multiple sclerosis, lupus, and Guillain-Barre syndrome. Individuals with other neurological disorders that are clinically mild and stable with medication, such as mild Parkinson's disease, will not be excluded.
11. Pregnant or lactating female.
12. Females planning to become pregnant or planning to discontinue contraceptive precautions within 60 days of enrollment in this study.
13. Any condition that in the opinion of the investigator would interfere with evaluation of the vaccine or interpretation of study results.
14. Participation in a novel A (H1N1) 2009 influenza vaccine study or a known history of novel A (H1N1) 2009 influenza infection.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4560 (Actual)
Dates: Start 2009-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of two injections of A (H1N1) 2009 influenza VLP vaccine | 35 days

SECONDARY OUTCOMES:
Evaluation of immunogenicity of two injections of A (H1N1) 2009 influenza VLP vaccine by Hemagglutination Inhibition | 35 days
Long-term Serious Adverse Events (SAEs) and Significant New Medical Conditions (SNMCs) | 6 months post second dose

CONTACTS AND LOCATIONS:
Overall Officials: Constantino R Lopez Macias, M.D., Principal Investigator — Specialities Hospital, National Medical Centre "Siglo XXI" Mexican Institute for Social Security (IMSS)
Locations (1):
- Specialities Hospital, National Medical Centre "Siglo XXI" Mexican Institute for Social Security (IMSS), Mexico City, Mexico